CLINICAL TRIAL: NCT04283994
Title: Using the Electronic Health Record to Identify and Promote Goals-of-Care Communication for Older Patients With Serious Illness
Brief Title: Project to Improve Communication About Serious Illness--Hospital Study: Comparative Effectiveness Trial (Trial 2)
Acronym: PICSI-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Erin Kross, Professor, Division of Pulmonary, Critical Care and Sleep Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00007031-B; 1R01AG006244 (NIH)
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Chronic Disease; Neoplasm Metastasis; Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure, Congestive; Liver Cirrhosis; Kidney Failure, Chronic; Lung Diseases, Interstitial; Peripheral Vascular Disease; Diabetes With End Organ Injury
Keywords: Patient care; Inpatients; Health Communication; Patient Care Planning; Quality of Life; Health care quality, access, and evaluation; Palliative care
MeSH Terms: conditions — Dementia; Chronic Disease; Neoplasm Metastasis; Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure; Liver Cirrhosis; Kidney Failure, Chronic; Lung Diseases, Interstitial; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Survey-based Patient/Clinician Jumpstart (Experimental): The Survey-based Patient/Clinician Jumpstart Guide will be developed with two types of data: 1) EHR data; and 2) Survey data. Using automated methods and NLP/ML algorithms, the presence/absence of POLST, advance directives and DPOA documentation will be identified from both inpatient and outpatient notes (e.g., progress notes, specialty consult notes, alerts and care plans) preceding the current hospitalization. The survey data will be completed by patients or their surrogate/family at enrollment and will provide assessments of the following: a) preferences for discussions about goals of care; b) most important barrier and facilitator for having such discussions; and c) current goals of care. These elements are contained within the Jumpstart guides and the information is tailored to each recipient (i.e., patient, surrogate/family, or clinician).
  Interventions: Behavioral: Survey-based Patient/Clinician Jumpstart
- EHR-based Clinician Jumpstart (Active Comparator): The EHR-based Clinician Jumpstart Guide will be developed by using automated methods and NLP/ML algorithms to both inpatient and outpatient EHR notes (e.g., progress notes, specialty consult notes, alerts and care plans) preceding the current hospitalization. It will summarize the presence/absence of POLST, advance directives and DPOA documentation. It will not include survey-based information.
  Interventions: Behavioral: EHR-based Clinician Jumpstart
- Usual care (No Intervention): Patients in this arm receive usual care; neither subjects nor providers will receive either version of the Jumpstart Guide.

INTERVENTIONS:
Behavioral: Survey-based Patient/Clinician Jumpstart — The Jumpstart Guide is a communication-priming intervention for clinicians, patients and their families that addresses hospitalized patients' goals of care. The intervention's goal is to prompt clinicians to provide standard of care which includes a discussion with patients or their legal surrogate decision-maker about their goals of care. The Jumpstart takes two forms. One is "EHR-based" and provides information to the clinician about prior advance care planning documentation derived from the EHR. The other is "bi-directional" and patient-specific (Survey-based Patient/Clinician Jumpstart Guide). It provides the same information as the EHR-based Clinician Jumpstart Guide but also includes information about patients' self-reported preferences for communication and care as well as primary barriers and facilitators to this communication. The Jumpstart Guides include tips to improve this communication for clinicians, patients and families.
  Other Names: Bidirectional Jumpstart Guide Intervention
  Arms: Survey-based Patient/Clinician Jumpstart
Behavioral: EHR-based Clinician Jumpstart — The Jumpstart Guide is a communication-priming intervention for clinicians that addresses hospitalized patients' goals of care. The intervention's goal is to prompt clinicians to provide standard of care which includes a discussion with patients or their legal surrogate decision-maker about their goals of care. The one-page EHR-based Clinician Jumpstart Guide provides information to the clinician about prior advance care planning documentation derived from the EHR. The EHR-based Clinician Jumpstart Guide includes tips to improve goals-of-care communication.
  Other Names: Clinician-facing Jumpstart Guide Intervention
  Arms: EHR-based Clinician Jumpstart

SUMMARY:
The objective of this protocol is to test the effectiveness of a Jumpstart intervention on patient-centered outcomes for patients with chronic illness by ensuring that they receive care that is concordant with their goals over time, and across settings and providers. This study is particularly interested in understanding the effect of the intervention to improve quality of palliative care for patients with Alzheimer's disease and related dementias (ADRD) but will also include other common chronic, life-limiting illnesses.

The specific aims are:

1. To evaluate the efficacy of the EHR-based clinician-facing Jumpstart, drawn from the electronic medical record (EHR), the survey-based bi-directional Jumpstart, drawn from patient or family completed surveys, and usual care for improving quality of care provided to patients with chronic illness experiencing a hospitalization. The primary outcome is EHR documentation of a goals-of-care discussion, assessed from randomization through 30 days. Secondary outcomes include: a) intensity of care outcomes (e.g., ICU use, ICU and hospital free days, hospital readmissions, costs of hospital care); and b) patient- and family-reported outcomes assessed by surveys at 3-5 days and 4-6 weeks after randomization, including occurrence and quality of goals-of-care discussions in the hospital, goal-concordant care, psychological symptoms, and quality of life.
2. To conduct a mixed-methods evaluation of the implementation of the interventions, guided by the RE-AIM and CFIR frameworks for implementation science, incorporating quantitative evaluation of the interventions' reach and adoption, as well as qualitative analyses of interviews with participants, to explore barriers and facilitators to future implementation and dissemination.

DETAILED DESCRIPTION:
OVERVIEW: Jumpstart is a communication-priming intervention for clinicians, patients and their families that focuses on hospitalized patients' goals of care. In this comparative effectiveness trial, the investigators examine the effectiveness of two approaches designed to promote goals-of-care discussions for older, seriously ill, hospitalized patients recruited from three UW Medicine hospitals. The two approaches include a survey-based bi-directional intervention and an EHR-based clinician-facing intervention. Both of these interventions provide clinicians with Jumpstart Guides that include data selected from the EHR on advance care planning as well as tips designed to improve communication about patients' goals of care and care preferences. Additionally, the survey-based bi-directional Jumpstart includes not only the EHR-based care planning information but also communication tips that are based on specific information from patients' (or surrogates) self-reported surveys. These bi-directional Jumpstarts are shared not only with clinicians but also with participating patients and families. The Jumpstart Guide is provided by email and in-person. This trial tests the comparative effectiveness of the survey-based bi-directional Jumpstart, the EHR-based clinician-facing Jumpstart and usual care. Unique to this trial is the use of the EHR to identify eligible participants, provide data for the intervention, and be the mechanism for delivering the intervention.

This current study is "Trial 2" of the R01 Award funding this trial. Trial 1 was completed prior to the initiation of Trial 2.

SPECIFIC AIM 1: Evaluate the effectiveness of the survey-based bi-directional Jumpstart compared to the EHR-based clinician-facing Jumpstart and usual care for improving quality of care.

TRIAL 2 has four components.

Component 1- Subject Identification/Recruitment/Randomization: Patients who meet the inclusion criteria are screened and identified using daily screening reports and staff review. The investigators oversample patients with ADRD to include 40% of the sample. Patients are approached by study staff in person during their hospital stay to assess their interest in participating in the study. Recruitment conversations are designed to take place in the patient's hospital room. Subjects are asked to complete surveys at three time points: 1) at enrollment; 2) 3-5 days after randomization; and 3) 4-6 weeks after randomization. Follow-up surveys may be completed in-person, by paper, online, or by phone, based on respondents' preferences.

If patients are not able to participate themselves (e.g., cognitive impairment, sedated or ventilated), the investigators recruit their legal surrogate decision-maker to participate. This surrogate (under Washington State Law RCW 7.70.065) provides consent on their own behalf and is a research study subject.

Eligible patients are assigned to one of the three interventions in a 1:1:1 ratio. Patients are randomized using variable size blocks and stratified for hospital and ADRD vs. no ADRD. Surrogates/families follow the randomization status of the patients whom they are representing.

Component 2- EHR-based clinician-facing Jumpstart guide: The Jumpstart guide is developed from an automated review of the EHR. It summarizes the presence/absence of POLST, advance directives and DPOA documentation. It provides general recommendations to assist clinicians in initiating goals of care discussions.

Component 3- Survey-based bi-directional Jumpstart Guide: Survey data, completed by patients or their surrogate/family at enrollment provide assessments of the following: a) preferences for discussions about goals of care; b) most important barrier and facilitator for having such discussions; and c) current goals of care. These elements are contained within the Jumpstart guides and the information is tailored to each recipient (i.e., patient, surrogate/family, or clinician). This version provides survey-response specific recommendations to initiate goals of care discussions.

Component 4- Delivery of the intervention:

Clinician delivery: Guides are delivered within the first few days (1-3) after randomization to the primary clinician team (attending and resident physicians and advanced practice providers) via secure email or in person. Study staff monitor the care team for the patient and ensure that any new providers also receive the Jumpstart guide.

Patient and family delivery: For the survey-based bi-directional Jumpstart arm, study staff provide the patient or surrogate with a version of the Jumpstart guide, tailored to be appropriate for patients or their surrogates (without information on EHR-based advance care planning documents) and following the same timeframe. Jumpstart guides are delivered to the patient or surrogate/family at the hospital.

Comparison group: We will compare all 3 arms (survey-based bi-directional Jumpstart, EHR-based clinician-facing Jumpstart, usual care) in three two-way comparisons.

Outcome Assessment: The primary outcome is EHR documentation of a goals-of-care discussion in the 30 days following randomization. All subjects are asked to complete questionnaires at enrollment. The questionnaires may be completed as computer-assisted interviews or on-line depending on the subject's preference. The study staff member enrolling the subjects notifies them of their randomization status at this time. Subjects randomized to the survey-based bi-directional Jumpstart arm complete additional questionnaire items used to create the Jumpstart Guide.

The research staff will contact all subjects in person (or by telephone or email) for the evaluation/post-intervention phase. Patient and surrogate/family subjects will complete surveys at 3-5 days and 4-6 weeks after randomization. Surveys can be completed by telephone, mail, or online; we will contact each patient or family/surrogate at each interval using their preferred modality. Subjects may complete the surveys with study staff in person (if the patient is still in the hospital), over the phone, online using REDCap, or on paper and return via mail. Surrogate/Family subjects will complete the same measures at the same intervals as patients with a few exceptions: families will complete the SF-1 for themselves as well as by proxy for patients.

Follow up contacts for subjects at 3-5 days follow-up will be as follows: If the patient is still hospitalized, in-person contact will be attempted (surrogates, who may not be reachable in person, may be contacted by their preferred mode); otherwise, contact will be attempted via phone, email, or mail per the subject's preference. Second and third contact attempts will be made using the subject's preferred mode 2 and 4 days later (7 and 14 days later for mail).

Follow-up contacts for subjects at 4-6 weeks follow-up will be as follows: initial contact by subject's preferred mode at 4 weeks from enrollment, followed by 4 additional contacts at an interval of every 4-7 days for phone and online, and an interval of every 7-10 days for mail. In all cases, only non-respondents will continue to be contacted.

For surrogates of patients who have died, after a minimum of 4 weeks following the patient death, an "after death" questionnaire will be sent to the subject using their preferred mode. The after-death questionnaire includes items related to treatment preferences, psychological distress (HADS), and health-related quality of life (SF1). The after-death questionnaire will be sent one time with no additional follow-ups.

At the end of study participation, study staff will collect additional information from the patient's electronic health record including intensity of care outcomes. Data will be abstracted using automated EHR data collection and "gold standard" manual abstraction using standardized methods for training and quality control.

Secondary outcomes also include the following patient- and surrogate/family-reported outcomes assessed by survey at 3-5 days and 4-6 weeks after randomization: occurrence and quality of goals-of-care communication in the hospital, goal concordant care, psychological symptoms, and quality of life.

SPECIFIC AIM 2: Evaluate the factors affecting the Jumpstart intervention implementation and identify barriers and facilitators to future implementation.

Patient and Surrogate/Family Subject Identification and Recruitment: Included in the patient's and surrogate/family member's consent form is a provision informing subjects that they may be contacted at the end of their study involvement to take part in a short, semi-structured interview to evaluate their study participation. Subjects will be sampled purposively to represent the following experiences: 1) participants from both intervention arms (EHR-based and survey-based); 2) participants who participated in the intervention fully as well as those who did not to better understand the reasons for less than full participation. "Full" participation is indicated by having completed all of the study materials.

Clinician Subject Identification and Recruitment: Study staff will recruit clinicians who were involved with the study to participate in a short interview after the clinician's study involvement with the enrolled patient has ended.

All interview participants will be selected using purposive sampling to ensure a diverse group (e.g., age, race/ethnicity, gender, specialty, year of training) in addition to the characteristics noted above.

Interview: Using an interview guide developed specifically for this project, interviewers will assess respondents' experience with the intervention and gather suggestions for ways to improve the intervention's content, delivery, and implementation, including implementation outcomes (e.g., acceptability, fidelity, penetration, maintenance) that will guide future dissemination of the intervention.

Assessment: Interviews are audio recorded, transcribed, and analyzed using thematic analysis. Validity and reliability are assessed by co-coding approaches.

ELIGIBILITY:
Eligibility criteria apply to three subject groups: 1) seriously ill adult patients; 2) adult surrogate legal next of kin of the patients; and 3) hospital clinicians.

Inclusion Criteria:

PATIENTS. Eligible patients will be those who are: 1) equal to or older than 80 years of age; or 2) equal to or older than 55 years of age with one or more chronic conditions used by the Dartmouth Atlas to study end-of-life care: malignant cancer/leukemia, chronic pulmonary disease, coronary artery disease, heart failure, chronic liver disease, chronic renal disease, dementia, diabetes with end-organ damage, and peripheral vascular disease, 3) English-speaking, 4) admitted for minimum of 12 hours/maximum of 96 hours to participating in-patient services at the participating hospitals, and 5) without documentation in the EHR of a goals-of-care discussion during this admission. Patients without decisional capacity (as documented in the EHR or as identified with a brief six-item screening tool) will be represented by a legal surrogate decision maker/legal next of kin (LNOK) in accordance with Washington State Law RCW 7.70.065.

SURROGATE/FAMILY. Eligible surrogate/family subjects will be those who are 18 years of age or older, English-speaking, involved in the patient's medical care or decision-making.

CLINICIANS (Interview). Eligible clinicians will be those who are 18 years of age or older, English-speaking, employed at a participating hospital, and have been the clinician of record for an enrolled patient in the trial.

Exclusion Criteria:

Reasons for exclusion for any patient in include: restricted status (prisoners or victims of violence); legal or risk management concerns (as determined by the attending physician or via hospital record designation); unable to complete informed consent procedures; and without a legal surrogate to participate for them. Patients who are non-English speaking (and therefore unable to complete survey materials) are excluded. Reasons for exclusion for any surrogate/family subject include: non-English speaking (and therefore unable to complete study materials), legal or risk management concerns (as determined by the attending physician or via hospital record designation); psychological illness or morbidity; and physical or mental limitations preventing ability to complete questionnaires. Patients under COVID precautions will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin K Kross, MD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Harborview Medical Center, Seattle, Washington
  - UW Medical Center - Northwest, Seattle, Washington
  - UW Medical Center - Montlake, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients and family/friend surrogates were screened and recruited from July 2021 to October 2023. Potential subjects were approached in the hospital by a research coordinator to assess interest and eligibility. Enrollees completed baseline surveys and were randomized. Patients and family were approached for interviews between December 2021 and May 2023. Clinicians were recruited for interviews in October 2020 (from Trial 1) and from January 2022 to May 2023 (from Trial 2).
Pre-assignment Details: 9262 patients were screened for eligibility, 6575 were excluded. 2687 patients/surrogates were approached for recruitment, 1563 were excluded as ineligible, 451 declined participation. Eligibility window expired for another 56 patient/surrogates. 617 subjects were enrolled and randomized for the primary outcome.
Groups:
- Survey-based Bi-directional Jumpstart [Patient]; EHR-based Clinician-facing Jumpstart [Patient]; Usual Care [Patient]: Patients: Randomized & completing follow-up assessments
- Survey-based Bi-directional Jumpstart [Family]; EHR-based Clinician-facing Jumpstart [Family]; Usual Care [Family]: Surrogate participants completing follow-up assessments
- Clinicians: Interview subjects only [T1/T2]
Period: Overall Study
Arm/Group | Survey-based Bi-directional Jumpstart [Patient] | EHR-based Clinician-facing Jumpstart [Patient] | Usual Care [Patient] | Survey-based Bi-directional Jumpstart [Family] | EHR-based Clinician-facing Jumpstart [Family] | Usual Care [Family] | Clinicians
Started | 203 | 205 | 209 | 33 | 36 | 40 | 30
Completed T2Q Survey [3-5 Days Post] | 99 | 112 | 118 | 23 | 23 | 28 | 0
Completed After-death (ADQ) Survey | 0 | 0 | 0 | 2 | 3 | 3 | 0
Completed T3Q Survey [4-6 Weeks Post] | 118 | 109 | 124 | 26 | 22 | 23 | 0
Completed Qualitative Interview | 8 | 2 | 0 | 5 | 0 | 0 | 0
Completed | 176 | 181 | 192 | 32 | 36 | 39 | 30
Not Completed | 27 | 24 | 17 | 1 | 0 | 1 | 0
Not completed — Death | 11 | 20 | 11 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 4 | 6 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patient data from medical records; family/friend surrogate data from self-report surveys. Clinician data from self-report at the time of interview.
Groups:
- Total: Total of all reporting groups
Arm/Group | Survey-based Bi-directional Jumpstart [Patient] | EHR-based Clinician-facing Jumpstart [Patient] | Usual Care [Patient] | Survey-based Bi-directional Jumpstart [Family] | EHR-based Clinician-facing Jumpstart [Family] | Usual Care [Family] | Clinicians | Total
Number analyzed (Participants) | 203 | 205 | 209 | 33 | 36 | 40 | 30 | 756
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 62 | 67 | 63 | 17 | 22 | 27 | 29 | 287
  >=65 years | 141 | 138 | 146 | 16 | 14 | 13 | 1 | 469
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [64.5 to 82] | 72 [63 to 80] | 71 [64 to 80] | 65 [57 to 75] | 61.5 [53.5 to 70] | 62 [55.75 to 67] | 38 [34.25 to 46] | 70 [62 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 94 | 92 | 15 | 26 | 25 | 16 | 355
  Male | 116 | 111 | 117 | 18 | 10 | 15 | 14 | 401
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 6 | 5 | 0 | 2 | 3 | 2 | 30
  Not Hispanic or Latino | 190 | 195 | 202 | 33 | 34 | 37 | 28 | 719
  Unknown or Not Reported | 1 | 4 | 2 | 0 | 0 | 0 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 8
  Asian | 5 | 11 | 7 | 0 | 4 | 1 | 5 | 33
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 6
  Black or African American | 12 | 17 | 15 | 2 | 2 | 1 | 0 | 49
  White | 175 | 163 | 177 | 31 | 28 | 32 | 24 | 630
  More than one race | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 7
  Unknown or Not Reported | 6 | 6 | 7 | 0 | 1 | 3 | 0 | 23
Region of Enrollment [Number; unit: participants]
  United States | 203 | 205 | 209 | 33 | 36 | 40 | 30 | 756
Diagnoses [Count of Participants; unit: Participants] — Collected from the patients' EHR. Eligibility diagnoses documented within the 2 years prior to randomization. Counts are not mutually exclusive and participants may have more than one categorical diagnosis. Population: Diagnoses were only collected for the 617 patient subjects.
  Participants
    dementia, confirmed via manual screening: number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    dementia, confirmed via manual screening | 24 | 25 | 28 |  |  |  |  | 77
    non-hematologic cancer: number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    non-hematologic cancer | 40 | 46 | 38 |  |  |  |  | 124
    hematologic cancer: number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    hematologic cancer | 2 | 0 | 7 |  |  |  |  | 9
    chronic obstructive pulmonary disease (COPD): number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    chronic obstructive pulmonary disease (COPD) | 46 | 46 | 49 |  |  |  |  | 141
    other chronic pulmonary disease: number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    other chronic pulmonary disease | 52 | 44 | 57 |  |  |  |  | 153
    coronary artery disease (CAD): number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    coronary artery disease (CAD) | 84 | 74 | 83 |  |  |  |  | 241
    congestive heart failure (CHF): number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    congestive heart failure (CHF) | 74 | 72 | 76 |  |  |  |  | 222
    peripheral vascular disease (PVD): number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    peripheral vascular disease (PVD) | 43 | 50 | 50 |  |  |  |  | 143
    liver disease: number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    liver disease | 31 | 27 | 23 |  |  |  |  | 81
    diabetes: number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    diabetes | 63 | 55 | 57 |  |  |  |  | 175
    renal disease: number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 0 | 617
    renal disease | 47 | 49 | 48 |  |  |  |  | 144
Hospital Site [Count of Participants; unit: Participants] — Collected from the electronic health record and institutional data. Population: Hospital site is only relevant for the 617 patient subjects who were randomized; and for the clinicians who worked at those locations.
  Participants
    number analyzed (Participants) | 203 | 205 | 209 | 0 | 0 | 0 | 30 | 647
    County [HMC] | 47 | 49 | 51 |  |  |  | 3 | 150
    University [UW-ML] | 81 | 81 | 82 |  |  |  | 7 | 251
    Community [UW-NW] | 75 | 75 | 76 |  |  |  | 7 | 233
    More than one location | 0 | 0 | 0 |  |  |  | 2 | 2
    Unknown/Not recorded | 0 | 0 | 0 |  |  |  | 11 | 11
Relationship to patient [Count of Participants; unit: Participants] — Relationship of the participating family member/friend to the patient subject, collected via self-report from Surrogate Survey Respondents Population: Relationship to patient was only relevant for the family/friend surrogates of the patients.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 33 | 36 | 40 | 0 | 109
    Spouse/partner |  |  |  | 12 | 9 | 9 |  | 30
    Adult child |  |  |  | 11 | 21 | 25 |  | 57
    Sibling |  |  |  | 6 | 3 | 3 |  | 12
    Parent |  |  |  | 0 | 0 | 0 |  | 0
    Other relative |  |  |  | 1 | 2 | 3 |  | 6
    Friend |  |  |  | 3 | 1 | 0 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: EHR Documentation of Goals of Care Discussions
Description: The primary outcome is the proportion of patients who have a goals-of-care discussion that has been documented in the electronic medical record (EHR) in the period between randomization and 30 days following randomization. The proportion is the number of patients with goals-of-care (GOC) documentation over the number of patients in each study arm. Documentation of goals-of-care discussions will be evaluated using our natural language processing/machine learning (NLP/ML) methods.
Time Frame: from randomization to 30 days post randomization
Population: All randomized participants
Measure: Number; unit: Proportion of participants
Groups:
- Survey Based Bi-directional Jumpstart Guide Intervention; EHR Based Clinician-facing Jumpstart Guide Intervention; Usual Care: No Intervention: Patient-or-LNOK-Proxy
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Proportion of participants | 0.271 | 0.317 | 0.206
Statistical Analysis 1: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; A total sample size of 600 (200 per arm) would give 80% power to detect a difference in proportions of 0.16 for each of the 3 pairwise comparisons assuming an overall 0.5 significance threshold, a Bonferroni adjustment for the 3 comparisons, and variance based on a proportion of 0.54; Test type: Superiority; p = 0.023, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.114, 95% CI 2-sided [0.030 to 0.197] — Risk difference = clinician-facing intervention - usual care. Estimated via linear regression after adjusting for hospital site and dementia diagnosis. Confidence intervals using robust standard errors
Statistical Analysis 2: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.294, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.068, 95% CI 2-sided [-0.013 to 0.150] — Risk difference = bidirectional intervention - usual care. Estimated via linear regression after adjusting for hospital site and dementia diagnosis. Confidence intervals using robust standard errors
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.952, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.045, 95% CI 2-sided [-0.134 to 0.044] — Risk difference = bidirectional intervention - clinician-facing intervention. Estimated via linear regression after adjusting for hospital site and dementia diagnosis. Confidence intervals using robust standard errors

2. Secondary Outcome: Intensity of Care: ICU Admissions (30 Days)
Description: Any new ICU admissions or readmissions collected from the EHR.
Time Frame: from randomization to 30 days post randomization
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Count of admissions per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Count of admissions per participant | 0.0887 (0.302) | 0.0634 (0.282) | 0.0622 (0.279)

3. Secondary Outcome: Intensity of Care: ICU Admissions (90 Days)
Description: Any new ICU admissions or readmissions collected from the EHR.
Time Frame: from randomization to 90 days post randomization
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Count of admissions per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Count of admissions per participant | 0.118 (0.367) | 0.117 (0.391) | 0.0957 (0.354)

4. Secondary Outcome: Intensity of Care: ICU Admissions (Post-discharge, 7 Days)
Description: Any ICU admissions or readmissions collected from the EHR. Censored at 90 days post-randomization.
Time Frame: 7-days post-discharge
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Count of admissions per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Count of admissions per participant | 0.015 (0.121) | 0.010 (0.099) | 0.000 (0.000)

5. Secondary Outcome: Intensity of Care: ICU Admissions (Post-discharge, 30 Days)
Description: Any ICU admissions or readmissions collected from the EHR. Censored at 90 days post-randomization.
Time Frame: 30-days post-discharge
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Count of admissions per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Count of admissions per participant | 0.030 (0.170) | 0.034 (0.207) | 0.024 (0.153)

6. Secondary Outcome: Intensity of Care: Hospital Readmissions (7 Days)
Description: Any hospital readmissions in 7 days following discharge; collected from the EHR. Censored at 90 days post-randomization.
Time Frame: readmissions in 7 days following discharge
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Count of admissions per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Count of admissions per participant | 0.0394 (0.195) | 0.0732 (0.261) | 0.0766 (0.267)

7. Secondary Outcome: Intensity of Care: Hospital Readmissions (30 Days)
Description: Any hospital readmissions in 30 days following discharge collected from the EHR. Censored at 90 days post-randomization.
Time Frame: readmissions in 30 days following discharge
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Count of admissions per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Count of admissions per participant | 0.128 (0.335) | 0.176 (0.463) | 0.230 (0.475)

8. Secondary Outcome: Intensity of Care: ICU Free Days (30 Days)
Description: Number of days alive and out of the ICU within 30 days from randomization, collected from the EHR.
Time Frame: from randomization to 30 days post randomization
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Number of days per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Number of days per participant | 28.1 (5.81) | 27.9 (6.17) | 28.5 (4.72)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 1.650, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.3 to 0.7] — Mean difference = bi-directional intervention - usual care. Estimated via linear regression after adjusting for hospital and dementia diagnosis. Confidence intervals using robust standard errors
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 0.985, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.6 to 0.5] — Mean difference = clinician-facing intervention - usual care. Estimated via linear regression after adjusting for hospital and dementia diagnosis. Confidence intervals using robust standard errors
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Test type: Superiority; p = 2.155, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.0 to 1.4] — Mean difference = bi-directional intervention - clinician-facing intervention. Estimated via linear regression after adjusting for hospital and dementia diagnosis. Confidence intervals using robust standard errors

9. Secondary Outcome: Intensity of Care: ICU Free Days (90 Days)
Description: Number of days alive and out of the ICU within 90 days from randomization, collected from the EHR.
Time Frame: from randomization to 90 days post randomization
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Number of days per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Number of days per participant | 83.8 (19.3) | 79.9 (24.3) | 83.1 (19.5)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 2.169, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis,; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-3.1 to 4.4] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 0.391, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-7.5 to 1.0] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Test type: Superiority; p = 0.210, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [-0.3 to 8.2] — [estimate comment as in outcome 8, analysis 3]

10. Secondary Outcome: Intensity of Care: Hospital Free Days (30 Days)
Description: Number of days alive and out of the hospital within 30 days from randomization; collected from the EHR.
Time Frame: from randomization to 30 days post randomization
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Number of days per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Number of days per participant | 21.6 (8.42) | 20.8 (9.16) | 20.8 (8.51)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 1.010, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.8 to 2.4] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 2.923, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-1.7 to 1.7] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Test type: Superiority; p = 1.034, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.9 to 2.5] — [estimate comment as in outcome 8, analysis 3]

11. Secondary Outcome: Intensity of Care: Hospital Free Days (90 Days)
Description: Number of days alive and out of the hospital within 90 days from randomization; collected from the EHR.
Time Frame: from randomization to 90 days post randomization
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Number of days per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Number of days per participant | 75.2 (21.6) | 70.5 (26.6) | 71.6 (24.4)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 0.384, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-1.0 to 7.9] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 1.923, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-6.1 to 3.7] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Test type: Superiority; p = 0.166, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [-0.1 to 9.4] — [estimate comment as in outcome 8, analysis 3]

12. Secondary Outcome: Patient or Surrogate/Family-reported Discussion of Goals (3-5 Days)
Description: Subjects will self-report (yes or no) if they had a discussion of goals of care ("the kind of medical care you/your loved one would want") during the index hospitalization. Responses of "unsure" are included in the sample and not counted as missing. This outcome is presented as a proportion: the number of participants reporting a goals-of-care discussion over the number of patients in each study arm.
Time Frame: 3-5 days after randomization
Population: Participants for which there is a response (potentially by a proxy) to this survey question. One response excluded as it was recorded as having occurred on day of randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 135 | 122 | 146
Participants | 48 | 39 | 62
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 0.160, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.11, 95% CI 2-sided [-0.23 to 0.00] — Risk difference = bi-directional intervention - usual care. Estimated via linear regression after adjusting for hospital and dementia diagnosis. Confidence intervals using robust standard errors
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 0.652, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.07, 95% CI 2-sided [-0.18 to 0.04] — Risk difference = clinician-facing intervention - usual care. Estimated via linear regression after adjusting for hospital and dementia diagnosis. Confidence intervals using robust standard errors
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 1.390, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.04, 95% CI 2-sided [-0.16 to 0.07] — Risk difference = bi-directional intervention - clinician-facing intervention. Estimated via linear regression after adjusting for hospital and dementia diagnosis. Confidence intervals using robust standard errors

13. Secondary Outcome: Patient or Surrogate/Family-reported Discussion of Goals (4-6 Weeks)
Description: Subjects will self-report (yes or no) if they had a discussion of goals of care ("the kind of medical care you/your loved one would want") during the index hospitalization. Responses of "unsure" are included in the sample and not counted as missing. This outcome is presented as a proportion: the number of subjects reporting a goals-of-care discussion over the number of patients in each study arm.
Time Frame: 4-6 weeks after randomization
Population: Participants for which there is a response (potentially by a proxy) to this survey question. Includes instances of proxies reporting on the measure after the death of a participant
Measure: Count of Participants; unit: Participants
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 144 | 132 | 150
Participants | 62 | 51 | 57
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 1.192, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.05, 95% CI 2-sided [-0.06 to 0.16] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 2.698, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.01, 95% CI 2-sided [-0.11 to 0.12] — [estimate comment as in outcome 12, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 1.477, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.08 to 0.16] — [estimate comment as in outcome 12, analysis 3]

14. Secondary Outcome: Quality of Communication (QOC)
Description: Quality of goals-of-care communication is assessed with the end-of-life communication scale (QOC_eol) of the Quality of Communication (QOC) survey. The QOC_eol subscale is based on 4 items, with item scores ranging from 0 (worst) to 10 (best). Responses of "My doctor has not done this" are converted into a rating of 0. Scores from the 4 items are summed together, resulting in a total score that ranges from 0 (worst) to 40 (best).
Time Frame: 3-5 days after randomization
Population: Participants for which there is a response (potentially by a proxy) which is numeric or can be converted to numeric for each of the 4 component questions. One response excluded as it was recorded as having occurred on day of randomization.
Measure: Mean (Standard Deviation); unit: Points on the scale
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 107 | 117 | 131
Points on the scale | 18.4 (14.4) | 18.4 (14.2) | 18.7 (14.7)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 2.293, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-4.30 to 3.16] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 2.381, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-4.11 to 3.14] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Test type: Superiority; p = 2.893, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-3.86 to 3.69] — [estimate comment as in outcome 8, analysis 3]

15. Secondary Outcome: SUPPORT Questions (3-5 Days)
Description: Concordance between the care patients want and the care they are receiving is measured with two questions from the SUPPORT study. The first defines patients' preferences: "If you/patient had to make a choice at this time, would you/they prefer a course of treatment focused on extending life as much as possible, even if it means having more pain and discomfort, or would you/they want a plan of care focused on relieving pain and discomfort as much as possible, even if that means not living as long?" The second question assesses perceptions of current treatment using the same two options. Responses of "unsure" are included in the sample and not counted as missing. The outcome is a dichotomous variable of whether the preference matches the report of care received.
Time Frame: 3-5 days after randomization
Population: Participants for which there is a response (potentially by a proxy) to both component questions. One response excluded as it was recorded as having occurred on day of randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 116 | 126 | 141
Participants | 46 | 64 | 56
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 2.829, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.00, 95% CI 2-sided [-0.13 to 0.12] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 0.188, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.11, 95% CI 2-sided [-0.01 to 0.24] — [estimate comment as in outcome 12, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 0.190, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.12, 95% CI 2-sided [-0.24 to 0.01] — [estimate comment as in outcome 12, analysis 3]

16. Secondary Outcome: SUPPORT Questions (4-6 Weeks)
Description: as for outcome 15
Time Frame: 4-6 weeks after randomization
Population: Participants for which there is a response (potentially by a proxy) to both component questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 134 | 123 | 143
Participants | 67 | 67 | 67
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 1.994, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.03, 95% CI 2-sided [-0.09 to 0.14] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 0.771, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.07, 95% CI 2-sided [-0.05 to 0.19] — [estimate comment as in outcome 12, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Complete case analysis. "Unsure" responses counted as non-events; Test type: Superiority; p = 1.447, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.04, 95% CI 2-sided [-0.17 to 0.08] — [estimate comment as in outcome 12, analysis 3]

17. Other Pre Specified Outcome: Intensity of Care: Palliative Care Consults Completed (30 Days)
Description: Any palliative care consults within 30-days post randomization
Time Frame: 30-days post randomization
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Count of consults per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Count of consults per participant | 0.0493 (0.217) | 0.0829 (0.279) | 0.0574 (0.271)

18. Other Pre Specified Outcome: Intensity of Care: Palliative Care Consults Completed (90 Days)
Description: Any palliative care consults within 90-days post randomization
Time Frame: 90-days post randomization
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Count of consults per participant
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Count of consults per participant | 0.0640 (0.245) | 0.107 (0.340) | 0.0670 (0.286)

19. Other Pre Specified Outcome: All-cause Mortality at 30 Days (Safety Outcome)
Description: From the electronic medical record and Washington State death certificates.
Time Frame: 30 days after randomization
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Participants | 11 | 18 | 14
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 1.836, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.012, 95% CI 2-sided [-0.058 to 0.034] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 1.250, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.021, 95% CI 2-sided [-0.030 to 0.073] — [estimate comment as in outcome 12, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Test type: Superiority; p = 0.581, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.033, 95% CI 2-sided [-0.084 to 0.017] — [estimate comment as in outcome 12, analysis 3]

20. Other Pre Specified Outcome: All-cause Mortality at 120 Days (Safety Outcome)
Description: From the electronic medical record and Washington State death certificates.
Time Frame: 120 days after randomization
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Participants | 21 | 37 | 30
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 0.692, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.039, 95% CI 2-sided [-0.102 to 0.025] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Test type: Superiority; p = 0.887, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = 0.038, 95% CI 2-sided [-0.033 to 0.109] — [estimate comment as in outcome 12, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Test type: Superiority; p = 0.080, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Risk Difference (RD) = -0.077, 95% CI 2-sided [-0.145 to -0.009] — [estimate comment as in outcome 12, analysis 3]

21. Other Pre Specified Outcome: Goals-of Care Discussions: Time to First Goals of Care Discussion
Description: Time to first goals of care discussion reported per person-day; collected from electronic health record. All participants contribute person-days until their death, the goals or care discussion, or 30 days post-randomization.
Time Frame: 30-days post randomization
Population: All participants contribute person-days until their death, the goals or care discussion, or 30 days post-randomization.
Measure: Number; unit: Incidence rate (per person-day)
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 203 | 205 | 209
Incidence rate (per person-day) | 0.0120 | 0.0147 | 0.0082
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Censoring by death; Test type: Superiority; p = 0.293, Regression, Cox — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test adjusting for hospital site and dementia diagnosis; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [0.9 to 2.1] — Hazard ratio = bi-directional intervention / usual care. Estimated via cox proportional hazards regression after adjusting for hospital and dementia diagnosis. Exponentiated Wald confidence intervals
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Censoring by death; Test type: Superiority; p = 0.027, Regression, Cox — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test adjusting for hospital site and dementia diagnosis; Hazard Ratio (HR) = 1.7, 95% CI 2-sided [1.1 to 2.5] — Hazard ratio = clinician-facing intervention / usual care. Estimated via cox proportional hazards regression after adjusting for hospital and dementia diagnosis. Exponentiated Wald confidence intervals
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Censoring by death; Test type: Superiority; p = 1.009, Regression, Cox — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test adjusting for hospital site and dementia diagnosis; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.6 to 1.2] — Hazard ratio = bi-directional intervention / clinician-facing intervention. Estimated via cox proportional hazards regression after adjusting for hospital and dementia diagnosis. Exponentiated Wald confidence intervals

22. Other Pre Specified Outcome: Anxiety (HADS Subscale)
Description: Symptoms of depression and anxiety assessed with the Hospital Anxiety and Depression Scale (HADS). The HADS is a reliable, valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress. Seven items evaluate anxiety. Each item is scored on a 4-point scale (ranging from 0-3) with scores for each subscale (anxiety and depression) ranging from 0-21. Higher scores reflect more symptoms of anxiety or depression.
Time Frame: 4-6 weeks after randomization
Population: Participants for which there is a response (all HADS questions asked about the person taking the survey, so no proxies could answer) which are numeric scores for each of the component questions.
Measure: Mean (Standard Deviation); unit: Points on the scale
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 107 | 102 | 115
Points on the scale | 5.79 (4.14) | 5.59 (4.25) | 6.20 (4.36)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 1.366, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.55 to 0.70] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 0.978, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.73 to 0.58] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Complete case analysis; Test type: Superiority; p = 2.390, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.99 to 1.30] — [estimate comment as in outcome 8, analysis 3]

23. Other Pre Specified Outcome: Depression (HADS Subscale)
Description: Symptoms of depression and anxiety assessed with the Hospital Anxiety and Depression Scale (HADS). The HADS is a reliable, valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress. Seven items evaluate depression. Each item is scored on a 4-point scale (ranging from 0-3) with scores for each subscale (anxiety and depression) ranging from 0-21. Higher scores reflect more symptoms of anxiety or depression.
Time Frame: 4-6 weeks after randomization
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Points on the scale
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 109 | 103 | 116
Points on the scale | 5.94 (4.05) | 6.32 (3.90) | 5.48 (3.81)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 1.125, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.57 to 1.51] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 0.258, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-0.13 to 1.94] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Complete case analysis; Test type: Superiority; p = 1.267, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.5 to 0.63] — [estimate comment as in outcome 8, analysis 3]

24. Other Pre Specified Outcome: EuroQol 5 Dimensions 5 Level (EQ-5D-5L)
Description: The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The 5 questions ask about problems with these domains, with response options on a 4-point Likert scale ranging from 1 (slight) to 4 (unable). Scores from the 5 questions are summed together, resulting in a total score ranging from 5 to 20. Higher scores reflect lower quality of life.
Time Frame: 4-6 weeks after randomization
Population: Participants for which there is a response (potentially by a proxy) which is numeric for each of the 5 component questions.
Measure: Mean (Standard Deviation); unit: Points on the scale
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 134 | 122 | 142
Points on the scale | 7.20 (4.23) | 7.11 (4.65) | 6.85 (4.66)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 1.594, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.68 to 1.32] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 1.803, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.79 to 1.36] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Complete case analysis; Test type: Superiority; p = 2.851, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-1.01 to 1.07] — [estimate comment as in outcome 8, analysis 3]

25. Other Pre Specified Outcome: CollaboRATE
Description: The CollaboRATE is patient- or proxy-reported measure of shared decision-making. This 3-question measure asks questions about how much effort was made by doctors and members of the healthcare team to help you understand your/their health issues, listen to what matters most to you/them about your/their health issues, and include what matters most to you/them in choosing what to do next. Answers range from 0 (no effort) to 4 (every effort). Scores from the 3 questions are summed together, resulting in a total score ranging from 0 (no effort) to 12 (highest effort). Higher scores reflect more engagement in shared decision-making.
Time Frame: 3-5 days after randomization
Population: Participants for which there is a numeric response (potentially by a proxy) for each of the 3 component questions. One response excluded as it was recorded as having occurred on day of randomization.
Measure: Mean (Standard Deviation); unit: Points on the scale
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 113 | 131 | 143
Points on the scale | 8.14 (2.87) | 8.16 (3.01) | 8.44 (2.66)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 1.243, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.97 to 0.40] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 1.032, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-1.00 to 0.35] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Complete case analysis; Test type: Superiority; p = 2.742, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.70 to 0.78] — [estimate comment as in outcome 8, analysis 3]

26. Other Pre Specified Outcome: Goal Concordance (3-5 Days)
Description: Concordance between the care patients want and the care they are receiving is measured by an investigator-developed question: "Do you think that your current medical care is in line with your goals?" Scale ranges from 0 (Not at all) to 4 (Completely). Higher scores reflect better goal-concordance.
Time Frame: 3-5 days after randomization
Population: Participants for which there is a numeric response (potentially by a proxy) for this survey question. One response excluded as it was recorded as having occurred on day of randomization.
Measure: Mean (Standard Deviation); unit: Points on the scale
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 119 | 130 | 141
Points on the scale | 3.05 (1.04) | 3.15 (0.881) | 3.06 (0.935)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 2.658, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.26 to 0.22] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 1.523, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.14 to 0.29] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Test type: Superiority; p = 1.381, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.33 to 0.15] — [estimate comment as in outcome 8, analysis 3]

27. Other Pre Specified Outcome: Goal Concordance (4-6 Weeks)
Description: as for outcome 26
Time Frame: 4-6 weeks after randomization
Population: Participants for which there is a numeric response (potentially by a proxy) for this survey question. Includes instances of proxies reporting on the measure after the death of a participant.
Measure: Mean (Standard Deviation); unit: Points on the scale
Arm/Group | Survey Based Bi-directional Jumpstart Guide Intervention | EHR Based Clinician-facing Jumpstart Guide Intervention | Usual Care: No Intervention
Number analyzed (Participants) | 139 | 131 | 146
Points on the scale | 3.06 (0.870) | 3.08 (0.977) | 3.03 (0.961)
Statistical Analysis 1: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 2.191, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.18 to 0.25] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: EHR Based Clinician-facing Jumpstart Guide Intervention vs Usual Care: No Intervention; Complete case analysis; Test type: Superiority; p = 2.138, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.19 to 0.27] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Survey Based Bi-directional Jumpstart Guide Intervention vs EHR Based Clinician-facing Jumpstart Guide Intervention; Complete case analysis; Test type: Superiority; p = 2.879, Regression, Linear — P-value is after a Bonferroni adjustment for three comparisons. The threshold for statistical significance was 0.05; Wald test with robust standard errors, adjusting for hospital site and dementia diagnosis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.23 to 022] — [estimate comment as in outcome 8, analysis 3]

ADVERSE EVENTS:
Time Frame: within 120 days of enrollment/randomization
Arm/Group | Survey-based Bi-directional Jumpstart [Patient] | EHR-based Clinician-facing Jumpstart [Patient] | Usual Care [Patient] | Survey-based Bi-directional Jumpstart [Family] | EHR-based Clinician-facing Jumpstart [Family] | Usual Care [Family] | Clinicians
All-Cause Mortality (participants affected / at risk) | 22/203 | 38/205 | 30/209 | 0/33 | 0/36 | 0/40 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/205 | 0/209 | 0/33 | 0/36 | 0/40 | 0/30
Other Adverse Events (participants affected / at risk) | 0/203 | 0/205 | 0/209 | 0/33 | 0/36 | 0/40 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04283994/Prot_SAP_001.pdf